CLINICAL TRIAL: NCT02323867
Title: UNRELATED AND PARTIALLY MATCHED RELATED DONOR PERIPHERAL STEM CELL TRANSPLANTATION WITH Alpha/Beta T CELL AND B CELL DEPLETION FOR PATIENTS WITH HEMATOLOGIC MALIGNANCIES
Brief Title: Allogeneic Stem Cell Transplant With Alpha/Beta T AND B Cell Depletion for Hematologic Malignancies
Acronym: AB-CliniMACs
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Timothy Olson, Medical Director, Hematopoietic Stem Cell Transplantation (HSCT) Program, Children's Hospital of Philadelphia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-010495; BT13BTθ51 (Other: The Children's Hospital of Philadelphia)
Record Dates: First submitted 2014-10-22; First posted 2014-12-24 (Estimated); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Leukemia; Lymphoma; Myelodysplasia
Keywords: Transplant; Alternative Donor
MeSH Terms: conditions — Leukemia; Lymphoma; Anemia, Refractory, with Excess of Blasts

STUDY DESIGN:
Intervention Model Description: intervention with device: Alpha Beta T cell depletion
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Alpha Beta Total Body Irradiation - total body irradiation (TBI) first (Experimental): Alpha Beta Total Body Irradiation - TBI first Day Treatment
  * 11 Anti-thymocyte globulin (ATG)
  * 10 ATG
  * 9 ATG
  * 8 TBI
  * 7 TBI
  * 6 TBI
  * 5 Thiotepa
  * 4 Thiotepa
  * 3 Cyclophosphamide
  * 2 Cyclophosphamide
  * 1 Rest 0 Transplant with alpha beta T cell depleted stem cells
- Alpha Beta Total Body Irradiation - TBI last (Experimental): Alpha Beta Total Body Irradiation - TBI last Day Treatment
  * 9 ATG
  * 8 ATG
  * 7 Thiotepa + ATG
  * 6 Thiotepa
  * 5 Cyclophosphamide
  * 4 Cyclophosphamide
  * 3 TBI
  * 2 TBI
  * 1 TBI 0 Transplant with alpha beta T cell depleted stem cells
- Alpha Beta Non-irradiation regimen (Experimental): Alpha Beta Non-irradiation regimen Day Treatment
  * 9 Busulfan + ATG
  * 8 Busulfan + ATG
  * 7 Busulfan +ATG
  * 6 Busulfan
  * 5 Thiotepa
  * 4 Thiotepa
  * 3 Cyclophosphamide
  * 2 Cyclophosphamide
  * 1 0 Transplant with alpha beta T cell depleted stem cells
  Interventions: Device: Alpha Beta T cell depletion

INTERVENTIONS:
Device: Alpha Beta T cell depletion
  Arms: Alpha Beta Non-irradiation regimen

SUMMARY:
This is a single arm pilot study for patients using α/β T cell-depleted peripheral Stem Cell Transplantation (PSCT) in with alternative donor sources with hematologic malignancies receiving alternative donor (unrelated or partially matched related) mobilized peripheral stem cells (PSCs) using the CliniMACS system for T cell depletion plus CD19+ B cell depletion to determine efficacy as determined by engraftment and graft versus host disease (GVHD), and one year leukemia free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Leukemias/lymphomas

   * Acute myeloid leukemia, primary or secondary Disease status: remission or <10% bone marrow blasts
   * Myelodysplasia
   * Acute lymphoblastic leukemia Disease status: in hematologic remission
   * Chronic myelogenous leukemia Disease status: chronic phase, accelerated phase or blast crisis now in second chronic phase.
   * Mixed lineage or biphenotypic acute leukemia
   * Lymphoblastic lymphoma Disease status: remission
   * Burkitt's lymphoma/leukemia: Disease status- in remission
2. Acceptable organ status clearance
3. No active untreated infection. Patients with possible fungal infections must have had at least 2 weeks of appropriate anti-fungal antibiotics and be asymptomatic
4. Signed informed consent.
5. Negative pregnancy test for females of childbearing potential.

Exclusion Criteria:

1. Patients who do not meet disease, organ or infectious criteria.
2. No suitable donor
3. Received previous allogeneic transplant

Donor must be either unrelated, mismatched up to one antigen/one antigen and one allele or a related, HLA match other than a sibling.

Max Age: 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-10; Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Engraftment: rates of engraftment, defined as the first day of Absolute Neutrophil Count (ANC) greater than 500 for the first of three consecutive days | 1 year

SECONDARY OUTCOMES:
Severe acute and chronic graft versus host disease (GVHD) | 1 year
  Estimation of the incidence and extent of acute and chronic GVHD. The overall incidence of acute GVHD, the incidence of Grade 4 acute GVHD and the incidence of chronic GVHD.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Olson, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Leahy AB, Li Y, Talano JA, Elgarten CW, Seif AE, Wang Y, Johnson B, Monos DS, Kadauke S, Olson TS, Freedman J, Wray L, Grupp SA, Bunin N. Unrelated donor alpha/beta T cell- and B cell-depleted HSCT for the treatment of pediatric acute leukemia. Blood Adv. 2022 Feb 22;6(4):1175-1185. doi: 10.1182/bloodadvances.2021005492. PMID 34872106